CLINICAL TRIAL: NCT06222710
Title: Pragmatic Randomized Controlled Trial of Ultrasound Guiding Pharmacopuncture Therapy for Supraspinatus Tendinopathy: a Pilot Study
Brief Title: Ultrasound Guiding Pharmacopuncture Therapy for Supraspinatus Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2023-04
Record Dates: First submitted 2023-12-22; First posted 2024-01-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pharmacological Action

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with ultrasound-guided pharmacoacupuncture (Experimental): 20 patients with ultrasound-guided pharmacoacupuncture
  Interventions: Procedure: Pharmacoacupuncture with ultrasound guiding
- Patients with blind pharmacoacupuncture (Active Comparator): 20 patients who treat pharmacoacupuncture without checking ultrasound images
  Interventions: Procedure: Pharmacoacupuncture without ultrasound guiding

INTERVENTIONS:
Procedure: Pharmacoacupuncture with ultrasound guiding — Physician choose the adequate type and dose of pharmacoacupuncture and needle type with ultrasound guiding
  Arms: Patients with ultrasound-guided pharmacoacupuncture
Procedure: Pharmacoacupuncture without ultrasound guiding — Physician choose the adequate type and dose of pharmacoacupuncture and needle type without ultrasound guiding
  Arms: Patients with blind pharmacoacupuncture

SUMMARY:
The purpose of this study is to confirm the comparative effect and accuracy of ultrasound procedures by conducting a practical randomized controlled clinical study comparing patients (20 patients) with ultrasound-guided pharmacoacupuncture and patients (20 patients) without checking ultrasound images in 40 patients with whom complain of moderate or higher pain with 5 or higher NRS when stabilizing the shoulder joint.

DETAILED DESCRIPTION:
This clinical study is conducted for the purpose of research, and it is a practical clinical study to confirm the comparative effect by comparing the strategy of treating patients with extreme myopathy (more than a month after the onset of symptoms) with ultrasound-guided acupuncture.

Supraspinatus tendonopathy is the most common of rotator cuff tendonopathy, which occurs most frequently among shoulder diseases. Inflammation of joints, muscles, and tendons often means tendinitis. Pain within a few days of acute manifestation can be diagnosed as tendinitis, but if it is older than a few months, degenerative changes in tissues may be the main cause rather than inflammation, and in this case, it is called tendinosis. Clinically, the line between tendinitis and tendinosis is unclear, and it is collectively referred to as tendinopathy because it is a series of successive pathological processes. Rotator cuff refers to the four muscles: hypertrophy, hypertrophy, distal, and subscapular muscles, which play the most important role in rotator cuff. About 95% of the muscles, when they lift their arms to the side or forward, regression occurs in the hypertrophy due to the anatomical structure, and it progresses to rupture when continuous regression or strong trauma occurs. Due to the anatomical characteristics, conservative treatment is strong in that the pain area is persistent and the risk of recurrence is high when the arm is moved.

Pharmacopuncture is a combination of acupuncture and drug therapy, which diagnoses a patient's constitution and disease condition and injects a certain amount of drugs extracted from specific herbal medicines into the treatment area to treat the disease. Ultrasound medical devices have the advantage of being able to perform high sensitivity, specificity, and dynamic tests, and being an inducer of not only diagnosis but also interventional treatment, allowing accurate procedures in real time without radiation exposure.

In this study, 40 patients with external pain in their shoulders and symptoms lasting more than a month will be assigned to 20 patients who are treated with ultrasound-guided acupuncture and 20 patients who are treated with acupuncture using tactile acupuncture. The recruitment of patients will be conducted in non-competitive recruitment and will be conducted until the recruitment of all patients (40 patients) is completed.

According to the schedule, patients will visit for a total of 12 treatments over a six-week period until the end of participation. After that, a total of two visits (weeks 7 and 13) will be made over a seven-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Those between 19 and 70 years of age.
* Those whose NRS (Numeric Rating Scale) of shoulder joint pain is 5 or higher and who complain of pain when abducting.
* When supraspinatus tendinopathy is confirmed on MRI.
* Those whose symptoms above last for more than 1 month.
* Those who agree to participate in clinical research and provide written test subject consent.

Exclusion Criteria:

* For patients diagnosed with a specific serious disease that may cause shoulder pain (acute fracture, dislocation of the shoulder, complete rupture of rotator cuff, etc.)
* For patients whose pain was caused by a condition other than the shoulder (tumor, fibromyalgia, rheumatoid arthritis, gout, cervical disc herniation, etc.)
* In patients with other chronic conditions (such as stroke and myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.) that may interfere with treatment effectiveness or interpretation of outcomes
* Patients currently taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect their findings
* Inadequate or unsafe medication: hemorrhagic disease, anticoagulant therapy, severe diabetic patients with risk of infection
* Patients who have taken drugs that can affect pain such as non-steroidal anti-inflammatory drugs (NSAIDs) within the last week or have experienced acupuncture treatment
* For patients who have received steroid injections within the last 3 months
* In the case of pregnant women and in the case of planning to become pregnant or nursing
* For patients within 6 months of shoulder surgery
* If it has not been one month since the end of participation in other clinical studies, or if you are planning to participate in other clinical studies within six months from the date of selection and participate in other clinical studies during the follow-up period
* If it is difficult to fill out a consent form to participate in the study
* In cases where it is difficult for other researchers to participate in clinical research

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain numeric rating scale, NRS | Week 1,2,3,4,5,6,7,13
  The intensity of spinal pain during the first week will be assessed using the NRS. In the NRS, patients choose a number from 0 to 10 that best describes their comfort (0 being no pain and 10 being the most comfortable they can imagine).

SECONDARY OUTCOMES:
Shoulder Pain And Disability Index, SPADI | Week 1,7,13
  The functional status of study subjects will be assessed using the SPADI questionnaire. SPADI is a 13-item questionnaire developed to assess the degree of disability related to shoulder pain. Each question is divided into 10 levels and consists of 5 questions in the pain evaluation section and 8 questions in the functional disability evaluation section. The higher the score, the more severe the disability. We will conduct an accredited Korean SPADI survey.
Range of motion, ROM | Week 1,2,3,4,5,6,7,13
  Active and passive ROM will be measured before and after treatment to evaluate the degree of improvement after treatment. ROM is evaluated by measuring the angle between the subject's upper limb and an imaginary line drawn vertically from the ground in the maximum range of motion of the subject's shoulder joint in flexion, extension, abduction, adduction, external rotation, and internal rotation. If measurement is not possible due to pain, it will be recorded as UC.
Neer test | Week 1,2,3,4,5,6,7,13
  Neer test is performed to evaluate the diagnostic significance before treatment and the degree of improvement after treatment. If measurement is not possible due to pain, it will be recorded as UC.
Empty can test | Week 1,2,3,4,5,6,7,13
  Empty can test is performed to evaluate the diagnostic significance before treatment and the degree of improvement after treatment. If measurement is not possible due to pain, it will be recorded as UC.
Full can test | Week 1,2,3,4,5,6,7,13
  Full can test is performed to evaluate the diagnostic significance before treatment and the degree of improvement after treatment. If measurement is not possible due to pain, it will be recorded as UC.
Hawkin's test | Week 1,2,3,4,5,6,7,13
  Hawkin's test is performed to evaluate the diagnostic significance before treatment and the degree of improvement after treatment. If measurement is not possible due to pain, it will be recorded as UC.
EuroQol-5 Dimension, EQ-5D-5L | Week 1,7,13
  EQ-5D-5L is a method of evaluating health status from various aspects and then indirectly calculating the quality weight of a specific health status using pre-assigned preference scores for each functional level. It is the most widely used among several indirect measurement methods. there is. The EQ-5D-5L consists of 5 questions. Each question includes mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Ask about the degree of depression, etc. Each item is weighted according to its level, and the preference score calculation equation is presented based on these weights and constants.
Patient Global Impression of Change, PGIC | Week 7,13
  This is a method that allows the patient to subjectively evaluate the degree of improvement on a 7-level scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Muscle test | Week 1,2,3,4,5,6,7,13
  To evaluate the degree of improvement in rotator cuff strength as shoulder stability is restored, the strength during external and internal rotation of the shoulder joint is compared with the healthy side. If measurement is not possible due to pain, it will be recorded as UC.

CONTACTS AND LOCATIONS:
Overall Officials: Sunah Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No